CLINICAL TRIAL: NCT04302961
Title: Effects of Gait Retraining With Auditory Feedback on Biomechanics and Ankle Joint Health in Individuals With Chronic Ankle Instability
Brief Title: Effects of Gait Retraining With Auditory Feedback
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: Principal Investigator, Luke Donovan, Assistant Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0552
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Ankle Injuries; Ankle Inversion Sprain
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory Feedback (Experimental): Participants will complete 8 sessions over a 2-week period of walking gait retraining on a treadmill while receiving auditory feedback.
  Interventions: Other: Auditory Feedback
- No Feedback (Active Comparator): Participants will complete 8 sessions over a 2-week period of walking on a treadmill without receiving feedback.
  Interventions: Other: No Feedback

INTERVENTIONS:
Other: Auditory Feedback — Participants will complete 8 sessions over a 2-week period of walking gait retraining on a treadmill while receiving no feedback. Participants will be instructed to walk on a treadmill at their desired pace in a manner that does not cause the auditory tool to elicit a noise.
  Arms: Auditory Feedback
Other: No Feedback — Participants will complete 8 sessions over a 2-week period of walking gait retraining on a treadmill while receiving no feedback. Participants will be instructed to walk on a treadmill at their desired pace in a manner that they perceive to be their normal walking speed and mechanics.
  Arms: No Feedback

SUMMARY:
There is evidence to support individuals with chronic ankle instability (CAI) have altered gait biomechanics which may lead to re-injury and poor patient outcomes. Currently, there are no interventions specifically targeting these abnormal gait biomechanics. Evidence supports the use of an external focus of attention feedback to promote motor learning and retention. The overall purpose of randomized clinical trial is to determine the effects of a 2-week (8 session) gait retraining protocol using an auditory external feedback instrument can (1) alter biomechanics during functional tasks (walking, step-down, lunge, lateral hops, and balance) (2) improve ankle cartilage measures and (3) improve patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one ankle sprain
* Index ankle sprain > 12 months prior to study enrollment
* Most recent ankle sprain > 12 weeks prior to study enrollment
* Score >10 on the Identification of Functional Ankle Instability (IdFAI) survey.
* Score <95% on the Foot and Ankle Ability Measure (FAAM) Activities of Daily Living and a <85% on the Sport subscales
* Be physically active by participating in some form of physical activity for at least 20 min per day, three times per week.

Exclusion Criteria:

* History of ankle surgery
* History of other musculoskeletal injuries within the past 6 weeks
* Any condition affecting plantar pressure distribution
* Neurological or vestibular disorders affecting balance
* Current/previous self-reported disability due to lower extremity pathology that may adversely affect neuromuscular function

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in lower extremity kinetics during walking | Immediate post-intervention, 1-week post-intervention
  Plantar pressure and center of pressure trajectory measured with an in-shoe plantar pressure system
Changes from baseline in talar cartilage deformation before and after walking | Immediate post-intervention, 1-week post-intervention
  Talar cartilage thickness and cross-sectional area will be measured with an diagnostic ultrasound imaging system
Changes from baseline in self-reported ankle function | Immediate post-intervention, 1-week post-intervention
  Changes from baseline in self-reported function as measured by the Foot and Ankle Ability Measure (FAAM) Activities of Daily Living and Sport questionnaire. Scores range from 100% (no decrease in function) to 0% (complete loss of function).

SECONDARY OUTCOMES:
Changes from baseline in static balance | Immediate post-intervention, 1-week post-intervention
  Static balance will be measured via a force plate
2. Changes from baseline in plantar pressure during forward lunges, lateral hops, and a step-down | Immediate post-intervention, 1-week post-intervention
  Plantar pressure during forward lunges, lateral hops, and a step-down will be recorded with an in-shoe insole system.

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torp DM, Thomas AC, Hubbard-Turner T, Donovan L. Plantar pressure profile during walking is associated with talar cartilage characteristics in individuals with chronic ankle instability. Clin Biomech (Bristol). 2022 May;95:105656. doi: 10.1016/j.clinbiomech.2022.105656. Epub 2022 Apr 27. PMID 35504121